CLINICAL TRIAL: NCT05264363
Title: Clinical Validation of the VIPUN GMS as a Gastric Motility Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIPUN Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LOTUS
Record Dates: First submitted 2022-02-10; First posted 2022-03-03 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Gastric Motor Function
Keywords: Medical device investigation

STUDY DESIGN:
Intervention Model Description: A prospective, interventional, single-arm, monocentric, investigation in a cohort of adult healthy subjects comprising a screening visit and a single study visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The main intervention is the application of the Investigational Medical Device (VIPUN Gastric Monitoring System prototype) together with the reference device (solid state high-resolution manometry) to record intraluminal pressure. The planned procedures are identical for all subjects in this single-arm investigation.
  Interventions: Device: VIPUN Gastric Monitoring System prototype

INTERVENTIONS:
Device: VIPUN Gastric Monitoring System prototype — The Investigational Medical Device (IMD) is used simultaneously with the reference device (solid state high-resolution manometry) to record gastric intraluminal pressure for approximately 2.5 hours.
  Other Names: VIPUN GMS

SUMMARY:
In order to validate that the VIPUN, Gastric Monitoring System (GMS) is a gastric motility monitoring system, we intend to show that the VIPUN GMS can assess motility through pressure measurement similar to high-resolution manometry (HRM).

In addition, the study aims to contribute to the design and development of a position confirmation functionality integrated in the VIPUN Gastric Monitoring System by establishing volume-pressure relations in the stomach and esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Aged between and including 18 and 65 years
* In good health on the basis of medical history and anamnesis by the Principal Investigator (or delegate)
* Agrees to refrain from drug, non-allowed medication, herbal supplement and dietary supplement intake on the day of the study visit
* Agrees to an overnight fast in advance of the study visit

Exclusion Criteria:

* Current or chronic gastrointestinal symptoms
* Use of any medication that might affect gastric function or visceral sensitivity in the opinion of the PI
* (Suspected) current use of illicit drugs
* Psychiatric or neurological illness
* Any history of gastrointestinal surgery that could influence normal gastric function in the opinion of the PI, including, but not limited to gastrectomy, esophagectomy, duodenotomy, pancreatectomy, bariatric surgery (bypass surgery, gastric banding…), placement of neuromodulator
* Simultaneous participation in other clinical studies
* Suspected or confirmed basal skull fracture, mid face trauma or maxillofacial trauma
* Nasopharyngeal surgery in the last 30 days
* History of severe coagulation abnormalities
* Therapeutic or prophylactic anticoagulation
* Gastrointestinal bleeding
* Ischemic bowel
* Peritonitis
* Deviated nasal septum impeding catheter placement
* Inability to pass a feeding tube through the nares (e.g. in case of anatomical features, nasal congestion or blockage)
* Recent (< 30 days) caustic ingestion (due to risk of esophageal rupture)
* Recent (< 30 days) esophageal varices (active, untreated or recently banded/cauterized)
* History of esophageal strictures
* History of gastric varices
* History of gastric obstruction
* History of gastrectomy, esophagectomy, duodeno-pancreatectomy, bypass surgery, gastric banding, bariatric balloon, or short bowel syndrome
* History of gastrostomy
* Allergy to components of the VIPUN Catheter
* Pregnancy or breastfeeding
* Allergy to components of the enteral nutrition
* Allergy to the available lubricants
* Allergy to the available local anesthetic
* Recent infection with SARS-CoV-2 (in the last 2 weeks prior to study visit).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Duration of gastric contractility on VIPUN GMS | protocol time T=0-120 minutes
  Time the smoothed and baseline-corrected VIPUN GMS pressure exceeds the contraction-threshold.
Duration of gastric contractility on manometry | protocol time T=0-120 minutes
  Time the smoothed and baseline-corrected gastric manometry pressure exceeds the contraction-threshold

SECONDARY OUTCOMES:
VIPUN GMS contraction frequency | protocol time T=0-120 minutes
  Gastric contractions identified visually by a expert gastroenterologists on the VIPUN GMS recording.
Manometry contraction frequency | protocol time T=0-120 minutes
  Gastric contractions identified visually by a expert gastroenterologists on the manometry recording.
Motility Tiled Runner contraction frequency | protocol time T=0-120 minutes
  Motility Tile Runner contractions are gastric contractions identified by the VIPUN Motility Tiled Runner software application.
Hallmarks of normal motility | protocol time T=0-150 minutes
  The presence/absence of hallmarks of normal gastric motility are scored by expert gastroenterologists on the VIPUN GMS pressure recording and on the manometry recording independently.
Duration of MMC phases | protocol time T=0-150 minutes
  The duration of MMC phase III is delineated by expert gastroenterologists on the VIPUN GMS pressure recording and on the manometry recording independently.
Nutrient-induced changes in tonic contractility | protocol time T=0-150 minutes
  Defined as the difference between baseline GMS pressure before and during nutrient administration.
Nutrient-induced changes in phasic contractility | protocol time T=0-150 minutes
  Defined as the difference between the frequency of Motility Tiled Runner contractions before and during nutrient administration.
Volume-pressure relation during stepwise inflation | Prior to protocol time T=0 minutes (=start motility recording).
  The pressure at each volume increment (range 0-135 ml) is recorded during stepwise inflation of the VIPUN GMS Catheter in the esophagus and in the stomach.

OTHER OUTCOMES:
Symptom severity | Throughout the study visit, specifically at baseline, during stepwise inflation (at each volume increment), and during the motility recording (at protocol time T=0, 60, 120 and 150 minutes).
  The severity of epigastric and nasopharyngeal symptoms are surveyed by means of a questionnaire throughout the study visit.
Device safety | Throughout study visit (from the moment the investigational medical device is applied until it is removed).
  All adverse events and device deficiencies are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, PhD, MD, Principal Investigator — KU Leuven
Locations (1):
- Translational Research Center for Gastrointestinal Disorders - KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No